CLINICAL TRIAL: NCT04274283
Title: A British Feasibility Study of Molecular Stratification and Targeted Therapy to Optimize the Clinical Management of Patients with Glioma by Enhancing Clinical Outcomes, Reducing Avoidable Toxicity, Improving Management of Post-operative Residual & Recurrent Disease and Improving Survivorship
Brief Title: Tessa Jowell BRAIN MATRIX - Platform Study
Acronym: BRAIN MATRIX
Status: Recruiting | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: The Brain Tumour Charity (Other); University of Oxford (Other); University of Edinburgh (Other); Genomics England (Unknown)
Responsible Party: Sponsor
Other Study IDs: RG_18-258; 14218060 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — * Fresh Frozen Tissue
  * Germline DNA
  * Liquid Biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Matched Tumour and Blood Sample - Research Pathway — For patient's undergoing surgery fresh tissue will be collected from the initial surgery and frozen until shipment to the Oxford BRAIN MATRIX Lab. Matched blood sample for germline DNA will be taken post-Platform Study entry. For patients with progression with available tumour samples from previous tumour surgery, blood will be collected and sent to Oxford along with their tumour samples.
  Samples will be shipped together to Oxford for molecular analysis (Whole Genome Sequencing (WGS) and EPIC array). The BRAIN MATRIX neuropathology and genomics team will produce an integrated report (histology, WGS, Heidelberg Classifier) for each case in consultation with the local neuropathology team. Once data is available, a virtual MDT with the BRAIN MATRIX neuropathology, genomics team and local site will be held to ensure all relevant information is incorporated in the final BRAIN MATRIX diagnostic report. The resulting integrated histological-molecular report will be available to local sites
Other: Matched Tumour and Blood Sample - NHS GMS pathway — Tessa Jowell BRAIN MATRIX centres in England can submit matched tissue and blood samples for Whole Genome Sequencing through the standard of care NHS Genomic Medicine Service pathway via their Genomic Laboratory Hub. For those from Devolved Nations, samples must go to the Oxford BRAIN MATRIX Laboratory who can facilitate the processing of samples through an alternative NHS GMS GLH or via the research pathway.

SUMMARY:
The main aim of the Tessa Jowell BRAIN MATRIX - Platform Study is to more precisely determine the exact type of tumour patients have by developing the essential infrastructure to provide rapid and accurate molecular diagnosis. A large network of clinical hubs across the United Kingdom, with expertise in managing patients with brain tumours, will be developed. Once established this infrastructure will facilitate the rapid introduction of clinical trials testing targeted therapies tailored to the genetic changes of an individual's tumour.

DETAILED DESCRIPTION:
Gliomas, a type of brain tumour, are the most common primary tumour of the central nervous system (CNS) and in 2016 there were 5250 deaths from brain tumours in the UK. However, brain tumours are a challenging disease to treat. The tumour's location within the brain and its tendency to grow into nearby brain tissue often make it very difficult to remove the tumour completely with surgery. There is also difficulty in delivering drugs in adequate amounts to the tumour due to the natural defences of the brain.

Brain tumours arise due to changes in the DNA and other molecules in cells of the brain. Different types of gliomas can have different changes and these can be used to determine a precise 'molecular diagnosis'. The ultimate goal for the Tessa Jowell BRAIN MATRIX is to learn how to use these molecular changes to more precisely determine what exact type of tumour patients have, and to identify, decide and test whether specific 'targeted' treatments could improve the survival and/or quality of life of patients with brain tumours.

Tessa Jowell BRAIN MATRIX is a programme of work, the principal purpose of which is to improve the knowledge of, and treatment for, glioma. The programme will include a Platform Study and subsequent interventional clinical trials. The Tessa Jowell BRAIN MATRIX Platform Study forms the backbone of this programme. In the Platform Study, the aim is to develop the infrastructure to provide rapid and accurate molecular diagnosis and the infrastructure to deliver clinical trials of new therapies in the future, thereby improving clinical outcomes in brain tumours.

The researchers aim to recruit 1,000 patients to the study. As gliomas occur at all ages and their specific subtype is hard to predict pre-operatively, the patient population eligible for the study is broad. A large network of clinical hubs across the UK, with expertise in managing patients with brain tumours, will be developed. Once established this infrastructure will facilitate the rapid introduction of clinical trials testing targeted therapies tailored to the genetic changes of an individual's tumour.

Eligible patients will either have had, or be about to have, surgery for their tumour. As part of this study, tumour removed during the operation will be analysed to look for specific molecular changes. As with normal standard care, the tumour will be analysed by a local pathologist. A small part will be sent for review by experts and advanced molecular analysis will be undertaken to get a detailed understanding of the DNA/molecular changes within the patient's tumour. These results will be fed back to the patient's treating doctor. It is intended that this will occur within 28 days; however, it may be longer while the study becomes fully operational.

If samples are available from a patient's previous surgery to their tumour, these may also be analysed. Similarly, if available, other relevant samples such as cerebrospinal fluid, collected as part of their care, may also be analysed. In addition, as technologies and analyses improve the understanding of brain tumours, the researchers may find important results at a later date. These will be fed back to the patient's doctor. Patients will also be asked to give a blood sample, which will also be analysed to look at the molecular features, including of their DNA. This is required to identify what 'new' changes have occurred in the patient's tumour. Following surgery, patients will continue with other treatment(s) as directed by their doctor.

Treatment generally involves radiotherapy and chemotherapy. As is standard practice, patients will be closely monitored for signs of disease progression and the effects of the treatment given. As part of this study, information on patients' treatments and disease will be collected.

Images from brain scans patients undergo, along with relevant clinical information, will also be sent to and stored by the University of Edinburgh, and where appropriate, undergo expert review by a panel of radiologists with expertise in brain tumours. If patients have further surgery, some of the tissue removed may also be analysed.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed suspected WHO Grade 2-4 glioma, (as evidenced radiologically) AND suitable for a diagnostic or therapeutic surgical procedure resulting in a tumour sample matched to a blood sample.
* Patients with progression with known WHO Grade 2-4 glioma (those with available frozen tumour will be prioritised for detailed genomic analysis).
* Valid written informed consent for the study.

Exclusion Criteria:

* Primary spinal cord tumours
* Active treatment of other malignancy
* Contraindication to MRI
* Patients without standard of care imaging available

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Patients with a newly diagnosed suspected WHO Grade 2-4 glioma, (as evidenced radiologically) AND suitable for a diagnostic or therapeutic surgical procedure resulting in a frozen tumour sample matched to a blood sample.
  * Patients with progression with known WHO Grade 2-4 glioma (those with available frozen tumour will be prioritised for detailed genomic analysis).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-24 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Time (from biopsy) to integrated histological-molecular diagnosis | 28 days
  This is defined as the difference (days) between date of biopsy and date of whole genome diagnosis and epigenomic classification.

SECONDARY OUTCOMES:
Time to completion of each node of tissue and imaging pathway | To be achieved within a timescale of up to 5 years
  The time to each node of the pathway will be measured from the date of receipt at the current node to date of delivery at the next.
Tumour and biological sample(s) quality control status | To be achieved within a timescale of up to 5 years
  Tumour and biological sample collection will be measured against protocol guidelines. These data will be collected in the surgical and pathological forms.
Imaging quality control status | To be achieved within a timescale of up to 5 years
  Imaging will be measured against established clinical guideline. The imaging form will measure compliance against these guidelines.
Inter-rater agreement of Response Assessment in Neuro-Oncology (RANO) | To be achieved within a timescale of up to 5 years
  Scans will be assessed and scored according to RANO criteria by the hub of Neuro-radiologists.
Extent of surgical resection | To be achieved within a timescale of up to 5 years
  Evaluated from the post-operative MRI scan and categorised as follows: Closed biopsy, open biopsy, debulking <50%, subtotal resection 50-90%, near total resection 90-<100%, gross total resection 100%.
Overall survival time | To be achieved within a timescale of up to 5 years
  Defined as the time from date of diagnosis to the date of death. Patients who are alive at the time of analysis will be censored at the date last seen in clinic.
Intracranial progression-free survival time | To be achieved within a timescale of up to 5 years
  Defined as the time from date of registration to the earliest of date of intracranial progressive disease or death from disease. The date of an event is defined as the earliest confirmation of progression by radiological assessment, clinical symptoms or MDT. Patients without progression at the time of analysis will be censored at the date last seen in clinic.
Quality of Life (QoL) scores | To be achieved within a timescale of up to 5 years
  Longitudinal measures of QoL will be generated from the QoL questionnaire according to the questionnaire-specific algorithm for scoring.
Type of interventions received | To be achieved within a timescale of up to 5 years
  Details of the type of interventions received will be monitored throughout the follow-up period and recorded on the Case Report Form.
Type of complications from treatments (standard of care) received. | To be achieved within a timescale of up to 5 years
  Details of complications relating to standard of care treatments received will be monitored throughout the follow-up period and recorded on the Case Report Form.
Concordance of diagnoses | To be achieved within a timescale of up to 5 years
  In relation to initial local radiological diagnosis, local pathological diagnosis and integrated histological-molecular diagnosis, any difference between the tiers of diagnoses will be highlighted and categorised as: discordant; agreed; refined.
Samples and images centrally stored | To be achieved within a timescale of up to 5 years
  Defined as confirmed central storage of images and material.
Targetable mutation(s) identified | To be achieved within a timescale of up to 5 years
  Relevant targetable mutations identified by Whole Genome Sequencing and Epigenomic Classification.
Post-mortem sampling consent status and sample collection confirmation | To be achieved within a timescale of up to 5 years
  Based on receipt of post-mortem consent form, and on post-mortem samples with confirmed central storage.
Number of applications to, and outputs resulting from data repository | To be achieved within a timescale of up to 5 years
  As per title.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Watts, Principal Investigator — Unviersity of Birmingham
Locations (13):
- United Kingdom (13):
  - Queen Elizabeth Hospital Birmingham, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Addenbrooke's Hospital, Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Lothian, Edinburgh
  - Queen Elizabeth Unviersity Hospital, NHS Greater Glasgow and Clyde Health Board, Glasgow
  - St James's University Hospital, Leeds Teaching Hospitals NHS Trust, Leeds
  - The Walton Centre, The Walton Centre NHS Foundation Trust, Liverpool
  - King's College Hospital, King's College Hospital NHS Foundation Trust, London
  - Charing Cross Hospital, Imperial College Healthcare NHS Trust, London
  - The Christie Hospital, The Christie NHS Foundation Trust, Manchester
  - Salford Royal Hospital, Northern Care Alliance NHS Foundation Trust, Manchester
  - Freeman Hospital, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Queen's Medical Centre, Nottingham University Hospitals NHS Trust, Nottingham
  - John Radcliffe Hospital, Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Scientifically sound proposals from appropriately qualified researchers will be considered for data sharing. Requests should be made by returning a Data Sharing Request Form to newbusiness@trials.bham.ac.uk; this captures the research requirements, statistical analysis plan, and intended publication schedule. Requests will be reviewed by the Cancer Research UK Clinical Trials Unit (CRCTU) Directors in discussion with the Chief Investigator (CI), Study Management Group (SMG) and independent Scientific Advisory Board (SAB). They will consider the scientific validity of the request, qualifications of the researchers, CI, SMG & SAB views, consent arrangements, practicality of anonymizing the requested data & contractual obligations. If supportive of the request, and where not already obtained, Sponsor consent for data transfer will be sought before notifying applicants of the outcome. It is anticipated that applicants will be notified within 3 months of receipt of the original request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be available within 1 year of study closure, if not before.
Access Criteria: See Plan Description above.

REFERENCES:
- [Background] Watts C, Savage J, Patel A, Mant R, Wykes V, Pohl U, Bulbeck H, Apps J, Sharpe R, Thompson G, Waldman AD, Ansorge O, Billingham L; TJBM Investigators. Protocol for the Tessa Jowell BRAIN MATRIX Platform Study. BMJ Open. 2022 Sep 8;12(9):e067123. doi: 10.1136/bmjopen-2022-067123. PMID 36378622
- See also: Trial Website — http://www.birmingham.ac.uk/research/crctu/trials/brain-matrix/index.aspx